CLINICAL TRIAL: NCT03035994
Title: Effect of Altered Mechanical Loading on Lower Extremity Biomechanics and Biochemical Markers in Individuals With an Anterior Cruciate Ligament Reconstruction
Brief Title: Effect of Altered Mechanical Loading in ACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-0409
Record Dates: First submitted 2017-01-22; First posted 2017-01-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Overloading (Experimental): Participants will walk on a force-instrumented treadmill for 20 minutes and will be provided visual biofeedback consisting of bilateral vertical ground reaction force. A target will be placed at 10% greater than the participant's baseline vertical ground reaction force. Participants will be asked to alter their walking gait in an attempt to reach the target line with each step.
  Interventions: Other: Real-Time Biofeedback
- Underloading (Experimental): Participants will walk on a force-instrumented treadmill for 20 minutes and will be provided visual biofeedback consisting of bilateral vertical ground reaction force. A target will be placed at 10% lower than the participant's baseline vertical ground reaction force. Participants will be asked to alter their walking gait in an attempt to reach the target line with each step.
  Interventions: Other: Real-Time Biofeedback
- Average (Experimental): Participants will walk on a force-instrumented treadmill for 20 minutes and will be provided visual biofeedback consisting of bilateral vertical ground reaction force. A target will be placed at the average of each participant's baseline vertical ground reaction force between limbs. Participants will be asked to alter their walking gait in an attempt to reach the target line with each step.
  Interventions: Other: Real-Time Biofeedback
- Control (No Intervention): Participants will walk for 20 minutes on a force-instrumented treadmill and will not be provided biofeedback.

INTERVENTIONS:
Other: Real-Time Biofeedback — A custom written MatLab script will sample bilateral peak vertical ground reaction forces and display the magnitude in real time on a screen placed in front of the participant. A target line will be placed in the middle of the screen which corresponds to one of the three loading conditions. Participants will be instructed to alter their movement in an attempt to match each limb's vertical ground reaction force to the target line.
  Arms: Average; Overloading; Underloading

SUMMARY:
Altered loading is a causative factor for the development of knee osteoarthritis following anterior cruciate ligament reconstruction (ACLR), and real-time biofeedback may be an effective intervention to manipulate altered mechanical loading about the knee. The purpose of this study is to 1) determine if ACLR participants are able to acquire and retain various loading patterns using real-time biofeedback, 2) determine the effect of altered loading on lower extremity biomechanics during walking gait, and 3) determine the effect of altered loading on biochemical markers of collagen turnover and inflammation during walking gait.

DETAILED DESCRIPTION:
Participants will attend 4 testing sessions. Lower extremity biomechanical outcomes and blood samples will be taken before and following the participant walking at a self-selected speed for 20 minutes. During the 20 minutes of treadmill walking real-time biofeedback will be displayed in an attempt to alter mechanical loading. Participants will complete a control, overloading, under-loading, average loading testing session. Order of loading condition will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of a primary, unilateral ACLR using either a hamstring or patellar tendon autograft, cleared by a physical for full return to physical activity with no limitations, and participate in at least 30 minutes of physical activity 3 times per week

Exclusion Criteria:

* History of injury to either leg, other than ACLR (e.g. ankle sprain, muscle strain), within 6 months prior to participation in the study, history of lower extremity surgery other than ACLR, history of osteoarthritis or current symptoms related to knee osteoarthritis (e.g. pain, swelling, stiffness), currently pregnant, or planning to become pregnant while enrolled in the study, cardiovascular restrictions that limit the participant's ability to participate in physical activity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Difference in acquisition as measured in root mean square error (RMSE) between loading conditions | Change in acquisition over 20 minute intervention
Difference in joint loading as measured in peak vertical ground reaction force normalized to body weight (xBW) between loading conditions | Change in joint loading over 20 minute intervention
Difference in cartilage turnover as measured in serum concentration of cartilage oligomeric matrix protein (pg/mL) between loading conditions | Chance in cartilage turnover over 20 minute intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luc-Harkey BA, Franz J, Hackney AC, Blackburn JT, Padua DA, Schwartz T, Davis-Wilson H, Spang J, Pietrosimone B. Immediate Biochemical Changes After Gait Biofeedback in Individuals With Anterior Cruciate Ligament Reconstruction. J Athl Train. 2020 Oct 1;55(10):1106-1115. doi: 10.4085/1062-6050-0372.19. PMID 32966563
- [Derived] Luc-Harkey BA, Franz JR, Blackburn JT, Padua DA, Hackney AC, Pietrosimone B. Real-time biofeedback can increase and decrease vertical ground reaction force, knee flexion excursion, and knee extension moment during walking in individuals with anterior cruciate ligament reconstruction. J Biomech. 2018 Jul 25;76:94-102. doi: 10.1016/j.jbiomech.2018.05.043. Epub 2018 Jun 15. PMID 29921523